CLINICAL TRIAL: NCT03477227
Title: Comparison of a Short Compression Hosiery (Stocking Without a Foot) With Standard Compression Stockings After Radiofrequency Ablation of Great Saphenous Vein With Phlebectomy: a Multicenter Randomized Controlled Non-inferiority Trial
Brief Title: New Compression Hosiery Versus Standard Class II Compression Stockings After Endothermal Ablation
Acronym: COSMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Collaborators: Medalp Private Surgery Clinic (Other); Research Clinical Centre of the Russian Railways, JSC (Other)
Responsible Party: Principal Investigator, Igor Zolotukhin, Clinical Professor, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COSMOS
Record Dates: First submitted 2018-03-15; First posted 2018-03-26 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Varicose Veins; Vascular Diseases
Keywords: compression stocking; elastic stocking; endovenous radiofrequency ablation; compression therapy
MeSH Terms: conditions — Varicose Veins; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short stocking (Experimental): After radiofrequency ablation of the GSF and phlebectomy varicose tributaries, patients will wear compression socks without foot for four weeks
  Interventions: Device: Short stocking
- Usual stocking (Active Comparator): After radiofrequency ablation of the GSF and phlebectomy varicose tributaries, patients will wear usual compression socks for four weeks (usual care)
  Interventions: Device: Usual stocking

INTERVENTIONS:
Device: Short stocking — Patients in the experimental group will be asked to wear new type of compression stockings for four weeks post-operatively
  Arms: Short stocking
Device: Usual stocking — Patients in the control group will be asked to wear usual type of compression 2 class stockings for four weeks post-operatively
  Arms: Usual stocking

SUMMARY:
A prospective comparative randomized multicentre non-inferiority trial. The purpose of this study is to compares of a short compression hosiery (stocking without a foot, compression class 2) with standard compression class 2 stockings for 7 days after the endovascular radiofrequency ablation of great saphenous vein with phlebectomy varicose tributaries.

DETAILED DESCRIPTION:
It is common practice to use compression hosiery in the postoperative period to reduce pain, swelling, ecchymosis and hematoms. Long-term compression therapy is associated with a number of inconveniences, which leads to a decrease in compliance and violation of the patient's appointed treatment schedule. The use of short compression stoking can improve the compliance to applying of compression in a round-the-clock mode while maintaining the effectiveness of therapy.

The aim of the study The purpose of this study is to compare a short compression hosiery (stocking without a foot, compression class 2) with standard compression class 2 stockings for 7 days after the endovascular radiofrequency ablation of great saphenous vein with phlebectomy varicose tributaries.

Materials and methods A Multicenter Randomized Controlled Non-inferiority Trial. The study compares the effectiveness of a short compression hosiery (stocking without a foot, compression class 2) with standard compression class 2 stockings for 7 days after the endovascular radiofrequency ablation of great saphenous vein with phlebectomy varicose tributaries.

The study includes patients who are scheduled for the radiofrequency ablation of the great saphenous vein and phlebectomy varicose tributaries (CEAP classification classes C2-C4).

Endpoints in the study: the main outcome (primary endpoint) is the quality of life according to CIVIQ questionnaire on the 30th day after the intervention. Additional outcomes (secondary endpoints): comfort of using short compression stocking with the visual analog scale (VAS), pain level with the visual analogue scale (VAS), foot swelling. Registration of results for additional outcomes is conducted on days 1, 7, 14 and 30.

The calculation of the sample size was made using the online calculator "Compare 2 Means: 2 Sample Non Inferiority or Superiority" (https://goo.gl/8ND8CQ). The sample size was calculated taking into account the average values for the CIVIQ quality of life questionnaire on day 30 after the endovascular treatment obtained by reviewing the literature. Selected parameters: first-order error (α) 2.5%; power 80%; boundaries of "non-inferiority limit" 5; the expected difference between the study groups of 0. Taking into account the possible dropout of patients from the study, the size of the groups is increased by 10%. The estimated sample size is 164 participants. Randomization of patients into groups is carried out with the help of the system of randomization of the site "Register of methods for treatment of chronic disease."

Statistical analysis. It is planned to conduct ITT - analysis (intentio-to-treat). For comparison, the primary and secondary outcomes will use nonparametric statistics (Mann-Whitney U-test).

Discussion The main purpose of this study is to evaluate the effectiveness of a new type of compression hosiery of a Russian manufacturer. The main hypotheses of the study: 1) it is expected that the absence of a "foot" in hosiery will increase the comfort of its use and increase the compliance of patients to the prescribed compression regime after intervention; 2) it is assumed that the lack of compression in the foot area will not lead to the development of its swelling and a decrease in the comfort of wearing compression hosiery.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age
* Symptomatic great saphenous vein (GSV) vein reflux > 0.5 seconds on color Duplex
* CEAP C2-C4 (inclusive)
* Informed consent

Exclusion Criteria:

* Symptomatic small saphenous vein (SSV) vein reflux
* CEAP Class C5 or C6 disease
* Prior GSV treatment
* History of deep vein thrombosis
* Acute deep or superficial vein thrombosis
* Pregnancy
* Patients who are unable to attend the hospital for follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2018-12-29 (Actual); Study Completion 2018-12-29 (Actual)

PRIMARY OUTCOMES:
Quality of life score measured by CIVIQ20 questionnaire | 30 days
  The specific quality of life score using the Chronic Venous Insufficiency Questionnaire (CIVIQ) score
  Calculation of the Global Index Score (GIS) of CIVIQ-20
  There are 20 questions in the CIVIQ-20, each with 5 possible answers (1 to 5), the minimum possible score being 20 and the maximum 100. In order to calculate the GIS, the difference between the final score and the minimum possible score is to be divided by the difference between the theoretical maximum and minimum scores (100-20=80), multiplied by 100.

SECONDARY OUTCOMES:
Pain level | 1, 7, 14, 21, 30 days
  Patient's post-procedure pain score using a visual analogue scale (VAS)
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
  The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Comfort of using compression hosiery | 1, 7, 14, 21, 30 days
  Comfort of using compression hosiery on a visual analogue scale (VAS)
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "comfort" anchor and the patient's mark, providing a range of scores from 0-100.
  The following cut points on the comfort VAS have been recommended: comfort (0-4 mm), mild comfort (5-44 mm), moderate comfort (45-74 mm), and no comfort (75-100 mm).

OTHER OUTCOMES:
Foot swelling | 1, 7, 14, 21, 30 days
  Circumference of the foot

CONTACTS AND LOCATIONS:
Overall Officials: Igor Zolotukhin, Principal Investigator — The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov
Locations (3):
- Russia (3):
  - The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov of the Ministry of health of the Russian Federation, Moscow
  - Road Clinical Hospital of JSC "Russian Railways", Saint Petersburg
  - Medalp Private Surgery Clinic, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Data collection will take place at the Russian Registry of Treatment of Chronic Venous Diseases (RRT CVD). Register in Russian. Registry now listed in the database ClinicalTrials.gov, ID NCT03035747 (see references)
Supporting Information: Study Protocol
Time Frame: Access to the data will be available after completion of the study.
Access Criteria: To access the data will need to send a request to RRT CVD administrator.
URL: http://www.venousregistry.org/index.php

REFERENCES:
- [Derived] Zolotukhin I, Demekhova M, Ilyukhin E, Sonkin I, Zakharova E, Efremova O, Kiseleva E, Gavrilov E. A randomized trial of class II compression sleeves for full legs versus stockings after thermal ablation with phlebectomy. J Vasc Surg Venous Lymphat Disord. 2021 Sep;9(5):1235-1240. doi: 10.1016/j.jvsv.2020.12.067. Epub 2021 Apr 20. PMID 33340729